CLINICAL TRIAL: NCT02512354
Title: Contribution of High-throughput Exome Sequencing in Fetopathology
Brief Title: Contribution of High-throughput Exome Sequencing in the Diagnosis of the Cause Fetal Polymalformation Syndromes
Acronym: FOETEX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: THEVENON PHRC I 2014
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Fetuses With at Least 2 Malformations, and no Diagnosis After Fetopathological and Radiological Examinations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fetus
  Interventions: Other: Sample of a fragment of fetal tissue; Other: Parent's blood samples

INTERVENTIONS:
Other: Sample of a fragment of fetal tissue
Other: Parent's blood samples

SUMMARY:
This research concerns the contribution of a new examination, high-throughput exome sequencing, in the diagnosis of the cause of polymalformative fetal syndromes. With currently available examinations, the causes of polyformative syndromes, which correspond to the association of several congenital malformations with varying degrees of severity in different organs, remain unknown in a large number of cases.

High-throughput exome sequencing (HTES) is a diagnostic tool that allows the simultaneous analysis of all of the coding parts of DNA. This examination has already shown its superior diagnostic capability in every post-natal diagnostic context, in particulier in infants with malformations associated or not with intellectual deficiency. Its contribution has not yet been studied in a large number of fetuses with polymalformations. To investigate the usefulness of HTES, we propose to carry out the examination in 100 fetuses with polymalformations, as well as the usual examinations including chromosomal microarray analysis and possibly the study of specific genes that may explain these malformations. A blood sample will be taken from both parents to allow interpretation of the results.

ELIGIBILITY:
Inclusion Criteria:

* Fetus with at least 2 malformations, with no diagnosis (or several low-certainty diagnostic hypotheses, which require several molecular examinations) after fetopathological and radiological examinations
* Written consent from both parents
* Possibility to obtain samples from both parents

Exclusion Criteria:

* Refusal of parents to take part in the study
* Parents without National Health Insurance cover
* Parents under guardianship or in custody
* Impossibility to obtain samples from both parents
* Diagnostic hypothesis considered highly probable for which a molecular test cheaper that HTES is available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fetuses With at Least 2 Malformations, and no Diagnosis After Fetopathological and Radiological Examinations
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Number of additional diagnoses made thanks to HTES compared with the usual examinations | baseline
Number of diagnoses not made by HTES compared with usual examinations | baseline

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de DIJON, Dijon
  - CHU Montpellier, Montpellier
  - CH de Mulhouse (Hôpital Emile Muller), Mulhouse
  - CHRU de Reims (Hôpital Maison Blanche), Reims
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de STRASBOURG (Hôpital Hautepierre), Strasbourg
  - CHRU de Tours, Tours
  - CHU de NANCY, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Lefebvre M, Bruel AL, Tisserant E, Bourgon N, Duffourd Y, Collardeau-Frachon S, Attie-Bitach T, Kuentz P, Assoum M, Schaefer E, El Chehadeh S, Antal MC, Kremer V, Girard-Lemaitre F, Mandel JL, Lehalle D, Nambot S, Jean-Marcais N, Houcinat N, Moutton S, Marle N, Lambert L, Jonveaux P, Foliguet B, Mazutti JP, Gaillard D, Alanio E, Poirisier C, Lebre AS, Aubert-Lenoir M, Arbez-Gindre F, Odent S, Quelin C, Loget P, Fradin M, Willems M, Bigi N, Perez MJ, Blesson S, Francannet C, Beaufrere AM, Patrier-Sallebert S, Guerrot AM, Goldenberg A, Brehin AC, Lespinasse J, Touraine R, Capri Y, Saint-Frison MH, Laurent N, Philippe C, Tran Mau-Them F, Thevenon J, Faivre L, Thauvin-Robinet C, Vitobello A. Genotype-first in a cohort of 95 fetuses with multiple congenital abnormalities: when exome sequencing reveals unexpected fetal phenotype-genotype correlations. J Med Genet. 2021 Jun;58(6):400-413. doi: 10.1136/jmedgenet-2020-106867. Epub 2020 Jul 30. PMID 32732226